CLINICAL TRIAL: NCT02807766
Title: Brain Plasticity of Autism in Response to Early Behavioral Intervention: A Multimodal MRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Huafu Chen, professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-chenhuafulab-001
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Autism
Keywords: autism; Brain Plasticity; Behavioral Intervention; Magnetic Resonance Imaging
MeSH Terms: conditions — Autistic Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sensory Integration Training (Experimental): Behavior modification and Sensory Integration Training
  Interventions: Behavioral: Behavior modification and sensory integration training
- applied behavioral analysis (Experimental): Behavior modification and applied behavioral analysis.
  Interventions: Behavioral: Behavior modification and applied behavioral analysis
- TEACCH (Experimental): Behavior modification and TEACCH.
  Interventions: Behavioral: Behavior modification and TEACCH
- Behavior modification (Other): Behavior modification.
  Interventions: Behavioral: Behavior modification
- healthy control group (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Behavior modification — Each group has 30 subjects and experiences six months' training.
  Arms: Behavior modification
Behavioral: Behavior modification and sensory integration training — Each group has 30 subjects and experiences six months' training.
  Arms: Sensory Integration Training
Behavioral: Behavior modification and applied behavioral analysis — Each group has 30 subjects and experiences six months' training.
  Arms: applied behavioral analysis
Behavioral: Behavior modification and TEACCH — Each group has 30 subjects and experiences six months' training.
  Arms: TEACCH

SUMMARY:
Autism is a well-recognized neurodevelopmental disorder severely affecting the health of children. While the unclear neurobiological basis of autism and the lack of effective medication, the most commonly used approach for treatment is behavioral intervention. However, the pathophysiological mechanisms underlying the intervention therapy remains incompletely understood. The current project aims to explore the impacts of different early behavioral intervention methods on brain plasticity of autism using multimodal MRI technique and provide guidelines for the intervention and treatment of autism by evaluating the efficiency of these methods.

DETAILED DESCRIPTION:
Autism is a well-recognized neurodevelopmental disorder severely affecting the health of children. While the unclear neurobiological basis of autism and the lack of effective medication, the most commonly used approach for treatment is behavioral intervention. However, the pathophysiological mechanisms underlying the intervention therapy remains incompletely understood. The current project aims to explore the impacts of different early behavioral intervention methods on brain plasticity of autism using multimodal MRI technique and provide guidelines for the intervention and treatment of autism by evaluating the efficiency of these methods. Investigators collect participants' brain imaging data, eye movement data, stool samples and clinical scale score before and after intervention. Investigators first investigate longitudinal effect of behavioral intervention on brain structure and function in children with autism. In addition, investigators provide new biological indexes upon multimodal large-scale brain connectomes to evaluate the curative effect of intervention. Finally, investigators propose a prediction model of intervention effect based on multimodal multivariate pattern analysis methods. Furthermore, investigators expect to map the state-of-the-art biomarkers on multi-modal networks to provide a new interpretation of pathophysiological mechanisms of autism.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 2 to 8 years old.
* Clinical DSM-IV diagnosis of autism.

Exclusion Criteria:

* Subjects with other neurodevelopmental diseases.
* Subjects with contraindications to MRI.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brain structural and functional change under behavioral intervention at 6 months in children with autism | through study completion, an average of 1 year
  Longitudinal effect of behavioral intervention on brain structure and function in children with autism will be assessed by Voxel-based morphometry analysis for structural changes, as well as Regional homogeneity, Amplitude of low-frequency fluctuation, etc, for functional changes.

SECONDARY OUTCOMES:
Prediction model of intervention effect based on multimodal multivariate pattern analysis methods | through study completion, an average of 1 year
  First, classify autism individuals into effective treatment group and ineffective treatment group according to the intervention effect at 6 months. Second, conduct feature selection with Sparse optimization algorithms and cluster analysis on MRI data. Third, design optimized classifiers integrated support vector machines and Gaussian Naive Bayes classifiers.

CONTACTS AND LOCATIONS:
Overall Officials: Huafu Chen, Principal Investigator — School of Life Science and Technology, University of Electronic Science and Technology of China
Locations (2):
- China (2):
  - Department of Children's and Adolescent Health, Public Health College of Harbin Medical University, Harbin, Heilongjiang
  - Center for Information in BioMedicine, Key laboratory for NeuroInformation of Ministry of Education, School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang X, Ming Y, Zhao W, Feng R, Zhou Y, Wu L, Wang J, Xiao J, Li L, Shan X, Cao J, Kang X, Chen H, Duan X. Developmental prediction modeling based on diffusion tensor imaging uncovering age-dependent heterogeneity in early childhood autistic brain. Mol Autism. 2023 Oct 30;14(1):41. doi: 10.1186/s13229-023-00573-2. PMID 37899464
- [Derived] Guo X, Duan X, Suckling J, Wang J, Kang X, Chen H, Biswal BB, Cao J, He C, Xiao J, Huang X, Wang R, Han S, Fan YS, Guo J, Zhao J, Wu L, Chen H. Mapping Progressive Gray Matter Alterations in Early Childhood Autistic Brain. Cereb Cortex. 2021 Feb 5;31(3):1500-1510. doi: 10.1093/cercor/bhaa304. PMID 33123725